CLINICAL TRIAL: NCT00135083
Title: One Versus Two Versus Three Daily Rapid-acting Insulin Injections of APIDRA (Insulin Glulisine) as add-on to Lantus® and Oral Sensitizer Basal Therapy in Type 2 Diabetes: a Multicenter, Randomized, Parallel, Open-label Clinical Study
Brief Title: Variable Bolus Regimen 1-2-3 for Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3511
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Once daily:
  * Insulin glulisine Dosing: Supper, Lunch, Breakfast
  * Monitoring Needed at: Bedtime,Pre-Supper, Pre-Lunch
  Interventions: Drug: insulin glulisine
- 2 (Experimental): Twice daily:
  * Insulin glulisine Dosing: Supper & Lunch, Lunch & Breakfast, Breakfast & Supper
  * Monitoring Needed at: Bedtime & Pre-Supper, Pre-Supper & Pre-Lunch, Pre-Lunch & Bedtime
  Interventions: Drug: insulin glulisine
- 3 (Experimental): Twice daily:
  * Insulin glulisine Dosing: Supper, Lunch, Breakfast
  * Monitoring Needed at: Bedtime, Pre-Supper, Pre-Lunch
  Interventions: Drug: insulin glulisine

INTERVENTIONS:
Drug: insulin glulisine — * Once Daily Insulin: Subjects will receive insulin glulisine administered once daily 0-15 minutes before the greatest glycemic impact meal of the day starting at one-tenth the total dose of insulin glargine with maximum starting dose of 10 Units, and with additional monitoring as shown in the table below.
  * Twice Daily: Subjects will receive insulin glulisine administered twice daily 0-15 minutes before the 2 greatest glycemic impact meals of the day starting at one-tenth the total dose of insulin glargine with a maximum starting dose of 10 Units, and with additional monitoring as shown in the table below.
  * Three Times Daily: Subjects will receive insulin glulisine administered 3 times daily 0-15 minutes before each meal of the day starting at one-tenth the total dose of insulin glargine with a maximum starting dose of 10 Units for each meal and additional monitoring as shown in the table below.

SUMMARY:
The purpose of this study is to show the non-inferiority of insulin glulisine administered with 1 meal versus 2 meals versus 3 daily meals, as measured by the change in hemoglobin A1c (HbA1c), from baseline to study week 24.

ELIGIBILITY:
Subjects with type 2 diabetes mellitus who have been using a stable combination oral antidiabetic therapy of 2 or 3 agents in different therapeutic classes for on at least 3 months will be enrolled in this study.

Inclusion Criteria:

* Male and female subjects 18 to 79 years of age with a diagnosis of type 2 diabetes mellitus for at least 6 months
* Current treatment with a stable dose of 2 oral antidiabetic agents. The oral agents must be in 2 or 3 of the following 3 different classes:

  * Sulfonylurea: dosage greater than or equal to, one-half the maximum recommended dosage (eg, glimepiride >/= 4 mg; glipizide, including gastrointestinal therapeutic system [GITS], >/= 10 mg; glyburide >/= 10 mg; Glynase® >/=3 mg). The dosage must have been stable for at least 3 months prior to screening.
  * Biguanide: metformin dosage ≥ 1000 mg daily, including Glucophage XR®. The dosage must have been stable for at least 3 months prior to screening.
  * Thiazolidinedione (TZD): pioglitazone >/= 15 mg or rosiglitazone >/= 24 mg. The subject must have been using the same thiazolidinedione for at least 6 months,and the dosage must have been stable for at least 3 months prior to screening.
* HbA1c >/= 8.0%
* Fasting C-peptide concentration > 0.27 nmol/L
* Able and willing to perform self-monitoring of blood glucose (SMBG) up to 4 times a day
* Able and willing to adhere to, and be compliant with, the study protocol
* Able to read English or Spanish at the sixth-grade level in order to complete the subject reported outcomes component of the study
* Signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

* Insulin use within the previous year
* History of hypoglycemia unawareness
* Acute or chronic, or history of, metabolic acidosis, including diabetic ketoacidosis
* Impaired renal function as shown by, but not limited to, serum creatinine ≥ 3mg/dL. For subjects taking metformin, serum creatinine >/= 1.5 mg/dL for males, or >/= 1.4 mg/dL for females.
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 2.5 times the upper limit of normal (ULN)
* Clinically significant peripheral edema if subject is using a TZD
* History of stroke, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, or angina pectoris, within the past 12 months
* History of, or current, congestive heart failure (New York Heart Association [NYHA] III-IV) requiring pharmacologic treatment
* Acute infection
* Any malignancy within the past 5 years, with the exception of adequately treated basal or squamous cell carcinoma or adequately treated cervical carcinoma in situ
* Current substance addiction or alcohol abuse or history of substance or alcohol abuse, within the past 2 years
* Any clinically significant renal disease (other than proteinuria) or hepatic disease
* Pregnant or lactating females
* Dementia or mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Impaired dexterity or vision rendering the subject unable to administer injections
* Known hypersensitivity to insulin glargine or insulin glulisine or any of the components of Lantus or Apidra
* Any disease or condition (including abuse of illicit drugs, prescription medications, or alcohol) that, in the opinion of the investigator or sponsor, may interfere with the completion of the study
* Unlikely to comply with the protocol, eg, uncooperative attitude, inability to return for follow-up visits, or unlikely to complete the study
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof, directly involved in the conduct of the protocol
* No subject will be allowed to enroll in this study more than once.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2004-08; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To show non-inferiority between treatment groups (insulin glargine plus insulin glulisine administered once a day, twice a day, or 3 times a day) in the change in glycemic control as measured by hemoglobin A1C. | From baseline to study week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barch, B.S., Study Director — Sanofi

REFERENCES:
- [Derived] Davidson MB, Raskin P, Tanenberg RJ, Vlajnic A, Hollander P. A stepwise approach to insulin therapy in patients with type 2 diabetes mellitus and basal insulin treatment failure. Endocr Pract. 2011 May-Jun;17(3):395-403. doi: 10.4158/EP10323.OR. PMID 21324825